CLINICAL TRIAL: NCT06137352
Title: Two Domestic HPV Vaccines (Wozehui ® and Cecolin ®) and Imported HPV Vaccines in Women Aged 13-14 Years Study on Immunogenicity：A Multi-center Cohort Study in China
Brief Title: Two Domestic HPV Vaccines and Imported HPV Vaccines in Women Aged 13-14 Years Study on Immunogenicity
Status: Not yet recruiting | Type: Observational
Sponsor: Fujian Maternity and Child Health Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HVAC2303
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: HPV Infection; HPV Vaccine; Cervical Cancer Prevention
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Venous Blood Samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescent females who received their first dose of HPV vaccine at 13-14 years: Adolescent females who completed their last dose of domestic bivalent HPV vaccine or imported HPV vaccine and were between 13 and 14 years of age at the time of the first dose. Two follow-up visits were conducted 12 months (window period ± 1 month) and 36 months (window period ± 1 month) after the last dose of vaccination.
  Interventions: Other: Follow up

INTERVENTIONS:
Other: Follow up — Each subject was recruited in 30-60 days after the last dose of domestic bivalent HPV vaccine or imported HPV vaccine, and followed up at 12 months (window period ± 1 month) and 36 months (window period ± 1 month) after the last dose of domestic bivalent HPV vaccine or imported HPV vaccine, with a total of two follow-up visits. At enrollment and both follow-up visits, subjects were required to collect 2 tubes of peripheral venous blood each.

SUMMARY:
This is a multi-center, open, prospective cohort study that aims to investigate the immunogenicity and immune persistence of two different domestically produced bivalent HPV vaccines compared with an imported HPV vaccine in women aged 13-14 years. A total of 3,000 subjects who have completed 2 doses of the domestic bivalent HPV vaccine and 3 doses of the imported HPV vaccine will be recruited from Fujian Maternal and Child Health Hospital as the initiator of the study, and will be recruited from a number of healthcare institutions nationwide. Of these, 1,000 subjects were vaccinated with the domestic bivalent HPV vaccine (Wozehui), 1,000 subjects were vaccinated with the domestic bivalent HPV vaccine (Cecolin), and 1,000 subjects were vaccinated with the imported HPV vaccine. Each subject was enrolled within 30-60 days after the last dose of domestic bivalent HPV vaccine or imported HPV vaccine, and a total of two follow-up visits were conducted 12 months (window period ± 1 month) and 36 months (window period ± 1 month) after the last dose of domestic bivalent HPV vaccine or imported HPV vaccine. In response to the WHO Cervical Cancer Elimination Strategy, domestic bivalent HPV vaccine has been offered free of charge to adolescent females aged 13-14 years, but there is still a lack of evidence comparing the antibody titer levels of domestic HPV vaccine and imported HPV vaccine in younger females. Therefore, we conducted the present immunogenicity study to explore the immunogenicity and immune persistence after vaccination with domestic bivalent HPV vaccine versus imported HPV vaccine in this age group of females.

DETAILED DESCRIPTION:
The study aims to: 1) Evaluate the immunogenicity of two different domestically produced bivalent HPV vaccines (Wozehui ® and Cecolin ®) versus imported HPV vaccines in adolescent females aged 13-14 years old; 2) Evaluate the immune persistence of two different domestically produced bivalent HPV vaccines (Wozehui ® and Cecolin ®) versus imported HPV vaccines in adolescent females aged 13-14 years old. This study is a multi-center, open, prospective cohort study with a total of 3,000 subjects recruited. According to the HPV vaccine that the participants received in the previous period, they were divided into 1,000 people in the domestic bivalent HPV vaccine group (Wozehui), 1,000 people in the domestic bivalent HPV vaccine group (Cecolin), and 1,000 people in the imported HPV vaccine group. Three immuneogenic blood was collected in all subjects 30-60 days, 12 months (window period ± 1 month) and 36 months (window period ± 1 month) after the last dose of either the domestic bivalent HPV vaccine or the imported HPV vaccine, which was used to perform HPV type 16 and 18 neutralizing antibody testing. The aim of this study was to evaluate the immunogenicity difference between two different domestically produced bivalent HPV vaccines and imported HPV vaccines in adolescent females aged 13-14 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have completed all procedures of domestic bivalent HPV vaccine or imported HPV vaccine and are 30-60 days from the last dose of vaccination at the time of enrollment;
* The participants are between 13-14 years old at the time of the first dose of domestic or imported HPV vaccination;
* The participant himself/herself and his/her guardian are able to provide proof of legal identity;
* The participant and his/her guardian are capable of understanding and signing the informed consent form;
* Participants are willing to complete study-related follow-up visits and blood collection as required by the protocol.

Exclusion Criteria:

* Participants who have received other marketed HPV vaccines, or who have participated in clinical studies of HPV vaccines, or who have participated in clinical studies of other vaccines within the last 6 months;
* Participants with congenital malformations, developmental disorders, genetic defects, and severe malnutrition that are severe or cause damage to vital organs;
* Participants with a history of epilepsy, psychosis, and major depression requiring medication, convulsions or seizures or a family history of psychosis;
* Participants who are immune compromised or have been diagnosed with congenital or acquired immunodeficiency, Human Immunodeficiency Virus (HIV) infection, lymphoma, leukemia, Systemic Lupus Erythematosus (SLE), Rheumatoid - - Arthritis, Juvenile Rheumatoid Arthritis (JRA), Inflammatory Bowel Disease (IBD), or other autoimmune disease, subjects who have received immunosuppressive therapy within the past 6 months;
* Absence of spleen, functional absence of spleen, and subjects with any condition resulting in absence of spleen or splenectomy;
* Subjects with physician-diagnosed coagulation abnormalities (e.g., coagulation factor deficiencies, coagulopathies, platelet abnormalities) or significant bruising or coagulation disorders;
* Participants who, in the judgment of the investigator, have any other factors that make them unsuitable for participation in a clinical trials.

Ages: 13 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescent females between the ages of 13-14 years old at the time of the first dose of HPV vaccination who have completed their last dose of domestic bivalent HPV vaccine or imported HPV vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The neutralization antibody GMT and antibody positivity testing at baseline | Baseline
  The neutralization antibody GMT and antibody positivity for HPV types 16 and 18 were tested
The neutralization antibody GMT and antibody positivity testing at 12-mouth follow-up | 12-month follow-up
  The neutralization antibody GMT and antibody positivity for HPV types 16 and 18 were tested 12 mouths after the last dose of domestic bivalent HPV vaccine or imported HPV vaccine.
The neutralization antibody GMT and antibody positivity testing at baseline 36-mouth follow-up | 36-month follow-up
  The neutralization antibody GMT and antibody positivity for HPV types 16 and 18 were tested 36 mouths after the last dose of domestic bivalent HPV vaccine or imported HPV vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Pengming Sun, Study Chair — Fujian Maternal and Child Health Hospital
Locations (1):
- Fujian Maternity and Child Health Hospital, Fuzhou, Fujian, China